CLINICAL TRIAL: NCT01288443
Title: A Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Study Evaluating the Efficacy and Safety of Five Doses and Two Dose Regimens of SAR236553 Over 12 Weeks in Patients With Primary Hypercholesterolemia and LDL-cholesterol ≥ 100 mg/dL (≥ 2.59 mmol/L) on Ongoing Stable Atorvastatin Therapy
Brief Title: Efficacy and Safety Evaluation of Alirocumab (SAR236553/REGN727) in Patients With Primary Hypercholesterolemia on Stable Atorvastatin Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFI11565; U1111-1116-5252 (Other: UTN)
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — alirocumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Placebo Q2W (Placebo Comparator): Placebo (for alirocumab) every 2 weeks (Q2W) for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Placebo (for alirocumab); Drug: Atorvastatin
- Alirocumab 50 mg Q2W (Experimental): Alirocumab 50 mg Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Alirocumab 100 mg Q2W (Experimental): Alirocumab 100 mg Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Alirocumab 150 mg Q2W (Experimental): Alirocumab 150 mg Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Alirocumab 200 mg Q4W (Experimental): Alirocumab 200 mg every 4 weeks (Q4W) and alternating placebo Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Placebo (for alirocumab); Drug: Atorvastatin
- Alirocumab 300 mg Q4W (Experimental): Alirocumab 300 mg Q4W and alternating placebo Q2W for 12-weeks in combination with atorvastatin stable dose.
  Interventions: Drug: Alirocumab; Drug: Placebo (for alirocumab); Drug: Atorvastatin

INTERVENTIONS:
Drug: Alirocumab — Two SC injections in the abdomen only.
  Other Names: SAR236553; REGN727
  Arms: Alirocumab 100 mg Q2W; Alirocumab 150 mg Q2W; Alirocumab 200 mg Q4W; Alirocumab 300 mg Q4W; Alirocumab 50 mg Q2W
Drug: Placebo (for alirocumab) — Two subcutaneous (SC) injections in the abdomen only.
  Arms: Alirocumab 200 mg Q4W; Alirocumab 300 mg Q4W; Placebo Q2W
Drug: Atorvastatin — Orally once daily at a stable dose of 10 mg, 20 mg, or 40 mg as background therapy.

SUMMARY:
Primary Objective:

* To evaluate the effect of alirocumab (SAR236553/REGN727) on low-density lipoprotein cholesterol (LDL-C) levels after 12 weeks of treatment in comparison with placebo in participants with LDL-C ≥ 100 mg/dL (≥ 2.59 mmol/L) on ongoing stable atorvastatin therapy.

Secondary Objectives:

* To evaluate the effects of alirocumab on other lipid levels after 12 weeks of treatment in comparison with placebo
* To evaluate the safety and tolerability of alirocumab
* To evaluate the development of anti-alirocumab antibodies
* To evaluate the pharmacokinetics of alirocumab

DETAILED DESCRIPTION:
The duration of study participation depended on the status of the participant at screening:

* For participants receiving atorvastatin 10 mg, 20 mg, or 40 mg at a stable dose for at least 6 weeks prior to screening, the study participation was to be approximately 21 weeks including a screening period of 1 week, a double-blind treatment period of 12 weeks and a follow-up period of 8 weeks.
* For participants receiving a lipid-lowering treatment other than atorvastatin or not at stable dose of atorvastatin 10 mg, 20 mg, or 40 mg for at least 6 weeks prior to screening, or drug naive participants, the study participation was to be approximately 27 weeks including a screening period of 1 week, a run-in treatment period with atorvastatin 10 mg, 20 mg, or 40 mg at a stable dose of 6 weeks, a double-blind treatment period of 12 weeks, and a follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* Participants with primary hypercholesterolemia receiving a lipid-lowering treatment other than atorvastatin or not at stable dose of atorvastatin 10 mg, 20 mg, or 40 mg for at least 6 weeks prior to screening period or drug naive participants if they are likely to have low-density lipoprotein cholesterol (LDL-C) ≥ 100 mg/dL (≥ 2.59 mmol/L) at the end of the 6-week run-in treatment period on atorvastatin therapy

OR

* Participants with primary hypercholesterolemia treated with atorvastatin at stable dose of 10 mg, 20 mg, or 40 mg for at least 6 weeks prior to screening period and likely to have LDL-C ≥ 100 mg/dL (≥ 2.59 mmol/L) at the screening visit

Exclusion criteria:

1. LDL-C < 100 mg/dL (< 2.59 mmol/L):

   * After the run-in period on atorvastatin (10 mg, 20 mg, or 40 mg) for participants receiving a lipid-lowering treatment other than atorvastatin or not at stable dose of atorvastatin 10 mg, 20 mg, or 40 mg for at least 6 weeks prior to the screening, or drug naive participant

   OR
   * At the first visit for participants who were being treated with stable dose of atorvastatin (10 mg, 20 mg, or 40 mg) for at least 6 weeks prior to screening
2. Participants not previously instructed on a cholesterol-lowering diet
3. Participants with type 1 diabetes
4. Participants with type 2 diabetes treated with insulin
5. Participants with type 2 diabetes and with an glycated hemoglobin (HbA1c) ≥ 8.5% at screening visit (considered poorly controlled)
6. Laboratory findings measured before randomization:

   * Triglycerides (TG) > 350 mg/dL (> 3.95 mmol/L) at screening visit
   * Positive serum or urine pregnancy test in females of childbearing potential
7. Pregnant or breast-feeding women
8. Women of childbearing potential with no effective contraceptive method

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (38):
- United States (38):
  - Investigational Site Number 840525, Tempe, Arizona
  - Investigational Site Number 840516, Los Angeles, California
  - Investigational Site Number 840528, Mission Viejo, California
  - Investigational Site Number 840509, Newport Beach, California
  - Investigational Site Number 840523, Palm Springs, California
  - Investigational Site Number 840534, Westlake Village, California
  - Investigational Site Number 840530, Colorado Springs, Colorado
  - Investigational Site Number 840504, Aventura, Florida
  - Investigational Site Number 840519, Aventura, Florida
  - Investigational Site Number 840514, Jacksonville, Florida
  - Investigational Site Number 840539, Jupiter, Florida
  - Investigational Site Number 840502, Miami, Florida
  - Investigational Site Number 840520, Pembroke Pines, Florida
  - Investigational Site Number 840524, Ponte Vedra, Florida
  - Investigational Site Number 840536, Port Orange, Florida
  - Investigational Site Number 840507, St. Petersburg, Florida
  - Investigational Site Number 840527, Chicago, Illinois
  - Investigational Site Number 840506, Evansville, Indiana
  - Investigational Site Number 840529, Indianapolis, Indiana
  - Investigational Site Number 840515, Wichita, Kansas
  - Investigational Site Number 840532, Madisonville, Kentucky
  - Investigational Site Number 840535, Auburn, Maine
  - Investigational Site Number 840503, Brockton, Massachusetts
  - Investigational Site Number 840512, Las Vegas, Nevada
  - Investigational Site Number 840505, Edison, New Jersey
  - Investigational Site Number 840538, Rochester, New York
  - Investigational Site Number 840508, Raleigh, North Carolina
  - Investigational Site Number 840522, Statesville, North Carolina
  - Investigational Site Number 840511, Cincinnati, Ohio
  - Investigational Site Number 840526, Cincinnati, Ohio
  - Investigational Site Number 840510, Lyndhurst, Ohio
  - Investigational Site Number 840533, Tulsa, Oklahoma
  - Investigational Site Number 840537, Eugene, Oregon
  - Investigational Site Number 840521, Bristol, Tennessee
  - Investigational Site Number 840531, Bountiful, Utah
  - Investigational Site Number 840517, Norfolk, Virginia
  - Investigational Site Number 840518, Richmond, Virginia
  - Investigational Site Number 840513, Olympia, Washington

REFERENCES:
- [Result] McKenney JM, Koren MJ, Kereiakes DJ, Hanotin C, Ferrand AC, Stein EA. Safety and efficacy of a monoclonal antibody to proprotein convertase subtilisin/kexin type 9 serine protease, SAR236553/REGN727, in patients with primary hypercholesterolemia receiving ongoing stable atorvastatin therapy. J Am Coll Cardiol. 2012 Jun 19;59(25):2344-53. doi: 10.1016/j.jacc.2012.03.007. Epub 2012 Mar 28. PMID 22463922
- [Result] Gaudet D, Kereiakes DJ, McKenney JM, Roth EM, Hanotin C, Gipe D, Du Y, Ferrand AC, Ginsberg HN, Stein EA. Effect of alirocumab, a monoclonal proprotein convertase subtilisin/kexin 9 antibody, on lipoprotein(a) concentrations (a pooled analysis of 150 mg every two weeks dosing from phase 2 trials). Am J Cardiol. 2014 Sep 1;114(5):711-5. doi: 10.1016/j.amjcard.2014.05.060. Epub 2014 Jun 18. PMID 25060413
- [Derived] Leiter LA, Tinahones FJ, Karalis DG, Bujas-Bobanovic M, Letierce A, Mandel J, Samuel R, Jones PH. Alirocumab safety in people with and without diabetes mellitus: pooled data from 14 ODYSSEY trials. Diabet Med. 2018 Dec;35(12):1742-1751. doi: 10.1111/dme.13817. Epub 2018 Oct 9. PMID 30183102
- [Derived] Toth PP, Hamon SC, Jones SR, Martin SS, Joshi PH, Kulkarni KR, Banerjee P, Hanotin C, Roth EM, McKenney JM. Effect of alirocumab on specific lipoprotein non-high-density lipoprotein cholesterol and subfractions as measured by the vertical auto profile method: analysis of 3 randomized trials versus placebo. Lipids Health Dis. 2016 Feb 13;15:28. doi: 10.1186/s12944-016-0197-4. PMID 26872608
- [Derived] Koren MJ, Kereiakes D, Pourfarzib R, Winegar D, Banerjee P, Hamon S, Hanotin C, McKenney JM. Effect of PCSK9 Inhibition by Alirocumab on Lipoprotein Particle Concentrations Determined by Nuclear Magnetic Resonance Spectroscopy. J Am Heart Assoc. 2015 Nov 19;4(11):e002224. doi: 10.1161/JAHA.115.002224. PMID 26586732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 38 centers in the United States of America. Overall, 514 participants were screened between January 2011 and August 2011, 331 of whom were screen failures and screen failures were mainly due to exclusion criteria met.
Pre-assignment Details: Randomization was stratified according to atorvastatin dose. Assignment to treatment arms was done centrally using an Interactive Voice/Web Response System in a 1:1:1:1:1:1 ratio after confirmation of selection criteria. 183 participants were randomized.
Groups:
- Placebo: Placebo (for alirocumab) every 2 weeks (Q2W) for 12-weeks in combination with atorvastatin stable dose.
- Alirocumab 200 mg Q4W: Alirocumab 200 mg every 4 weeks (Q4W) and alternating placebo (for alirocumab) Q2W for 12-weeks in combination with atorvastatin stable dose.
- Alirocumab 300 mg Q4W: Alirocumab 300 mg Q4W and alternating placebo (for alirocumab) Q2W for 12-weeks in combination with atorvastatin stable dose.
Period: Overall Study
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Started | 31 (Randomized) | 30 (Randomized) | 31 (Randomized) | 31 (Randomized) | 30 (Randomized) | 30 (Randomized)
Treated | 31 | 30 | 31 | 31 | 29 | 30
Completed | 31 | 29 | 30 | 27 | 23 | 25
Not Completed | 0 | 1 | 1 | 4 | 7 | 5
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 3 | 1
Not completed — Poor compliance to protocol | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Moved | 0 | 0 | 0 | 1 | 2 | 1
Not completed — Consent withdrawn by Participant | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Study drug auto-injector administration | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other than above | 0 | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population.
Groups:
- Placebo: Placebo (for alirocumab) Q2W for 12-weeks in combination with atorvastatin stable dose.
- Alirocumab 200 mg Q4W: Alirocumab 200 mg Q4W and alternating placebo (for alirocumab) Q2W for 12-weeks in combination with atorvastatin stable dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W | Total
Number analyzed (Participants) | 31 | 30 | 31 | 31 | 30 | 30 | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (8.5) | 58.5 (9.1) | 58.1 (9.2) | 59.9 (11.1) | 54.9 (10.8) | 55.5 (10.1) | 56.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 18 | 21 | 13 | 16 | 96
  Male | 16 | 17 | 13 | 10 | 17 | 14 | 87
Low-Density Lipoprotein Cholesterol (LDL-C) in mmol/L [Mean (Standard Deviation); unit: mmol/L] — Number of participants analysed = 31, 30, 31, 31, 29, 30 and 182, respectively.
  mmol/L | 3.4 (0.7) | 3.2 (0.7) | 3.3 (0.8) | 3.2 (0.7) | 3.3 (0.5) | 3.4 (0.6) | 3.3 (0.7)
LDL-C in mg/dL [Mean (Standard Deviation); unit: mg/dL] — Number of participants analysed = 31, 30, 31, 31, 29, 30 and 182, respectively.
  mg/dL | 130.2 (27.3) | 123.2 (27.9) | 127.0 (30.4) | 124.7 (26.9) | 127.2 (19.6) | 131.6 (24.8) | 127.3 (26.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Calculated LDL-C at Week 12 - On-Treatment Analysis
Description: Calculated LDL-C values were obtained using the Friedewald formula. Baseline adjusted least squares (LS) means and standard errors were estimated using an analysis of covariance (ANCOVA) model including available post-baseline data on treatment from first study drug injection up to 21 days after last study drug injection (on-treatment analysis). Missing Week 12 data were imputed by last observation carried forward [LOCF] method.
Time Frame: Baseline to Week 12 (LOCF)
Population: Modified Intent-To-Treat (mITT) population included all randomized participants with one baseline and at least one post baseline on-treatment calculated LDL-C.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 31 | 30 | 31 | 29 | 28 | 30
percent change | -5.1 (3.1) | -39.6 (3.2) | -64.2 (3.1) | -72.4 (3.2) | -43.2 (3.3) | -47.7 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Alirocumab 150 mg Q2W; Each treatment group was compared to placebo using ANCOVA-derived contrasts. A hierarchical testing procedure was applied to ensure strong control of overall Type-I error rate at 0.05 level. Order was following: 1. Alirocumab 150 mg Q2W versus placebo 2. Alirocumab 300 mg Q4W versus placebo 3. Alirocumab 100 mg Q2W versus placebo 4. Alirocumab 200 mg Q4W versus placebo 5. Alirocumab 50 mg Q2W versus placebo Testing continued only when high-order test was statistically significant at 5% level; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤ 0.05
Statistical Analysis 2: Comparison: Placebo vs Alirocumab 300 mg Q4W; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤ 0.05
Statistical Analysis 3: Comparison: Placebo vs Alirocumab 100 mg Q2W; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤ 0.05
Statistical Analysis 4: Comparison: Placebo vs Alirocumab 200 mg Q4W; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤ 0.05
Statistical Analysis 5: Comparison: Placebo vs Alirocumab 50 mg Q2W; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance ≤ 0.05

2. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mmol/L) at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 31 | 30 | 31 | 29 | 28 | 30
mmol/L | -0.20 (0.10) | -1.37 (0.10) | -2.10 (0.10) | -2.38 (0.10) | -1.46 (0.11) | -1.62 (0.10)

3. Secondary Outcome: Absolute Change From Baseline in Calculated LDL-C (mg/dL) at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: mITT population.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 31 | 30 | 31 | 29 | 28 | 30
mg/dL | -7.6 (3.9) | -53.0 (4.0) | -81.2 (3.9) | -92.0 (4.0) | -56.4 (4.1) | -62.5 (4.0)

4. Secondary Outcome: Percentage of Participants Achieving Calculated LDL-C <100 mg/dL (2.59 mmol/L) and <70 mg/dL (1.81 mmol/L) at Week 12 - On-Treatment Analysis
Time Frame: Week 12 (LOCF)
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 31 | 30 | 31 | 29 | 28 | 30
percentage of participants
  LDL-C <100 mg/dL (2.59 mmol/L) | 16.1 | 93.3 | 96.8 | 100.0 | 89.3 | 96.7
  LDL-C <70 mg/dL (1.81 mmol/L) | 3.2 | 46.7 | 83.9 | 100.0 | 46.4 | 56.7

5. Secondary Outcome: Percent Change From Baseline in Total Cholesterol, High-density Lipoprotein Cholesterol (HDL-C), Non-HDL-C and Apolipoprotein B (Apo-B) at Week 12 - On-Treatment Analysis
Description: Adjusted LS means and standard errors were estimated using the same ANCOVA model as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post-baseline on-treatment value for lipid parameters analyzed. Here, n signifies the number of participants analysed for each lipid parameter.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 31 | 30 | 31 | 29 | 28 | 30
percent change
  Total Cholesterol (n= 31, 30, 31, 29, 28, 30) | -1.6 (2.3) | -23.0 (2.3) | -39.7 (2.3) | -45.2 (2.3) | -28.0 (2.4) | -29.8 (2.3)
  HDL-C (n= 31, 30, 31, 29, 28, 30) | -1.0 (2.3) | 6.7 (2.4) | 4.1 (2.3) | 5.5 (2.4) | 6.3 (2.5) | 8.5 (2.4)
  Non-HDL-C (n= 31, 30, 31, 29, 28, 30) | -2.2 (2.9) | -33.6 (2.9) | -55.6 (2.9) | -62.5 (3.0) | -37.4 (3.0) | -40.7 (2.9)
  Apo-B (n= 30, 30, 30, 29, 27, 30) | 2.2 (2.9) | -27.3 (2.9) | -48.1 (2.9) | -56.1 (2.9) | -28.7 (3.1) | -33.1 (2.9)

6. Secondary Outcome: Percent Change From Baseline in Fasting Triglycerides and Lipoprotein(a) at Week 12 - On-Treatment Analysis
Description: Since the assumptions of normal distribution and equality of variances were not verified for the lipid parameters, percent changes were expressed as median (inter-quartile range).
Time Frame: Baseline to Week 12 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post-baseline on-treatment value for lipid parameters analyzed. Here, n signifies number of participants analysed for each lipid parameter.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 31 | 30 | 31 | 29 | 28 | 30
percent change
  Fasting Triglycerides (n= 31, 30, 31, 29, 28, 30) | 9.7 [-15 to 30.7] | -6.6 [-17.7 to 7.1] | -5.5 [-22.1 to 10.7] | -18.9 [-31.7 to -6.1] | -10.8 [-25.4 to 13.3] | -8.4 [-21.5 to 10.1]
  Lipoprotein(a) (n= 30, 30, 30, 29, 27, 30) | 0.0 [-11.8 to 11.5] | -13.3 [-33.3 to 0.0] | -26.1 [-36.7 to -8.0] | -28.6 [-46.9 to -22.2] | -16.7 [-33.3 to -6.3] | -7.9 [-18.8 to 0.0]

7. Secondary Outcome: Absolute Change in the Ratio Apolipoprotein B/Apolipoprotein A-1 (ApoB/ApoA-1) From Baseline to Week 12 - On-Treatment Analysis
Description: Adjusted LS mean and standard errors were estimated using the same ANCOVA as for primary endpoint.
Time Frame: Baseline to Week 12 (LOCF)
Population: Participants of the mITT population with one baseline and at least one post-baseline on-treatment value for ApoB/ApoA-1 ratio analyzed.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Number analyzed (Participants) | 30 | 30 | 30 | 29 | 27 | 30
ratio | 0.05 (0.03) | -0.23 (0.03) | -0.35 (0.03) | -0.42 (0.03) | -0.23 (0.03) | -0.29 (0.03)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 20) regardless of seriousness or relationship to investigational medicinal product (IMP).
Description: AEs that developed/worsened during 'treatment emergent period' (from 1st dose to last dose of IMP+70 days) are reported. Safety population:participants who received at least 1 dose or partial dose of IMP. 2 participants in 300 mg Q4W group received at least 1 dose of 150 mg and as per pre-specified algorithm they were included in 200 mg Q4W group.
Arm/Group | Placebo | Alirocumab 50 mg Q2W | Alirocumab 100 mg Q2W | Alirocumab 150 mg Q2W | Alirocumab 200 mg Q4W | Alirocumab 300 mg Q4W
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/30 | 1/31 | 0/31 | 1/31 | 1/28
Other Adverse Events (participants affected / at risk) | 10/31 | 14/30 | 14/31 | 12/31 | 12/31 | 10/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Alirocumab 50 mg Q2W (N=30) | Alirocumab 100 mg Q2W (N=31) | Alirocumab 150 mg Q2W (N=31) | Alirocumab 200 mg Q4W (N=31) | Alirocumab 300 mg Q4W (N=28)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=31) | Alirocumab 50 mg Q2W (N=30) | Alirocumab 100 mg Q2W (N=31) | Alirocumab 150 mg Q2W (N=31) | Alirocumab 200 mg Q4W (N=31) | Alirocumab 300 mg Q4W (N=28)
Sinusitis (Infections and infestations) | 3 | 0 | 1 | 2 | 1 | 0
Influenza (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 3 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 2 | 1 | 1 | 1
Bundle branch block left (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 2
Injection site erythema (General disorders) | 0 | 0 | 3 | 3 | 1 | 1
Injection site pruritus (General disorders) | 0 | 0 | 2 | 3 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 2 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 1 | 2 | 1 | 0
Injection site haematoma (General disorders) | 0 | 2 | 1 | 1 | 0 | 0
Injection site rash (General disorders) | 0 | 2 | 0 | 1 | 1 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 1 | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 2
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.